CLINICAL TRIAL: NCT02477644
Title: Randomized, Double-Blind, Phase III Trial Olaparib vs. Placebo Patients With Advanced FIGO Stage IIIB-IV High Grade Serious or Endometrioid Ovarian, Fallopian Tube, or Peritoneal Cancer Treated Standard First-Line Treatment
Brief Title: Platine, Avastin and OLAparib in 1st Line
Acronym: PAOLA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcagy Research (Other)
Collaborators: Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom Germany (Other); Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); Grupo Español de Investigación en Cáncer de Ovario (Other); Belgian Gynaecological Oncology Group (Other); Multicenter Italian Trials in Ovarian cancer and gynecologic malignancies (Unknown); Mario Negri Gynecologic Oncology group (MaNGO) (Other); Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other); Gynecologic Oncology Trial & Investigation Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GINECO-OV125b
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
Keywords: Advanced FIGO IIIB; IV high grade serious ovarian cancer; endometrioid ovarian cancer; standard first-line treatment; platinum-taxane chemotherapy; bevacizumab; olaparib; placebo
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib (Experimental): Tablets per os 300 mg
  Interventions: Drug: Olaparib
- Placebo (Placebo Comparator): Tablets per os 300 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olaparib — Tablets, per os, 300 mg twice daily;
  Arms: Olaparib
Drug: Placebo — Tablets, per os, 300 mg twice daily.
  Arms: Placebo

SUMMARY:
Randomized, Double-Blind, Phase III Trial of Olaparib vs. Placebo in Patients with Advanced FIGO Stage IIIB - IV High Grade Serous or Endometrioid Ovarian, Fallopian Tube, or Peritoneal Cancer treated with standard First-Line Treatment, Combining Platinum-Taxane Chemotherapy and Bevacizumab Concurrent with Chemotherapy and in Maintenance.

DETAILED DESCRIPTION:
Patients with advanced FIGO stage IIIB - IV high grade serous or endometrioid ovarian, fallopian tube, or peritoneal cancer treated with standard first-line treatment, combining platinum-taxane chemotherapy and bevacizumab concurrent with chemotherapy and in maintenance.

ELIGIBILITY:
Inclusion Criteria:

I-1. Female Patient must be ≥18 years of age. I-2. Signed informed consent and ability to comply with treatment and follow-up.

I-3. Patient with newly diagnosed I-3-1 Ovarian cancer, primary peritoneal cancer and/or fallopian-tube cancer,

I-3-2 Histologically confirmed (based on local histopathological findings):

* high grade serous or
* high grade endometrioid or
* other epithelial non mucinous ovarian cancer in a patient with germline BRCA 1 or 2 deleterious mutation I-3-3 at an advanced stage: FIGO stage IIIB, IIIC, or IV of the 1988 FIGO classification.

I-4. Patient who has completed prior to randomization first line platinum-taxane chemotherapy:

1. Platinum-taxane based regimen must have consisted of a minimum of 6 treatment cycles and a maximum of 9. However if platinum based therapy must be discontinued early as a result of non hematological toxicity specifically related to the platinum regimen, (i.e. neurotoxicity, hypersensitivity etc.), patient must have received a minimum of 4 cycles of the platinum regimen.
2. Intravenous, intraperitoneal, or neoadjuvant platinum based chemotherapy is allowed; for weekly therapy, three weeks are considered one cycle. Interval debulking is allowed.

I-5. Patient must have received prior to randomization a minimum of 3 cycles of bevacizumab in combination with the 3 last cycles of platinum-based chemotherapy. Only in case of interval debulking surgery, it is allowed to realize only 2 cycles of bevacizumab in combination with the last 3 cycles of platinium-based chemotherapy. Bevacizumab treatment should be administered at a dose 15mg/kg q3 weeks up to a total of 15 months.

I-6. Patient must be prior to randomization without evidence of disease (NED) or in complete response (CR) or partial response (PR) from her first line treatment. There should be no clinical evidence of disease progression (physical exam, imagery, CA 125) throughout her first line treatment and prior to study randomization.

I-7. Patient must be randomized at least 3 weeks and no more than 9 weeks after her last dose of chemotherapy (last dose is the day of the last infusion) and all major toxicities from the previous chemotherapy must have resolved to CTC AE grade 1 or better (except alopecia and peripheral neuropathy).

I-8. Patient must have normal organ and bone marrow function:

1. Hemoglobin ≥ 10.0 g/dL.
2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
3. Platelet count ≥ 100 x 109/L.
4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
5. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN.
6. Serum creatinine ≤ 1.25 x institutional ULN and creatinine clearance > 50 mL/min.
7. Patient not receiving anticoagulant medication who has an International Normalized Ratio (INR) ≤1.5 and an Activated ProThrombin Time (aPTT) ≤1.5 x ULN.

   The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or APTT is within therapeutic limits (according to site medical standard). If the patient is on oral anticoagulants, dose has to be stable for at least two weeks at the time of randomization.
8. Urine dipstick for proteinuria < 2+. If urine dipstick i s ≥2+, 24-hour urine must demonstrate <1 g of protein in 24 hours.
9. Normal blood pressure or adequately treated and controlled hypertension (systolic BP ≤ 140 mmHg and/or diastolic BP ≤ 90 mmHg).

I-9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1. I-10. Formalin fixed, paraffin embedded (FFPE) tumor sample from the primary cancer must be available for central BRCA testing and test result must be available for stratification.

I-11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment. (see appendix 4) I-12. For France only: In France, a subject will be eligible for randomization in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

E-1. Non-epithelial origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors).

E-2. Ovarian tumors of low malignant potential (e.g. borderline tumors), or mucinous carcinoma.

E-3. Patient with synchronous primary endometrial cancer unless both of the following criteria are met:

1. stage < II,
2. Less than 60 years old at the time of diagnosis of endometrial cancer with stage IA or IB grade 1 or 2, or stage IA grade III endometrioid adenocarcinoma OR ≥ 60 years old at the time of diagnosis of endometrial cancer with stage IA grade 1 or 2 endometrioid adenocarcinoma.

Patient with serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium is not eligible.

E-4. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS). Patient with a history of localized malignancy diagnosed over 5 years ago may be eligible provided she completed her adjuvant systemic therapy prior to randomization and that the patient remains free of recurrent or metastatic disease.

Patient with history of primary triple negative breast cancer may be eligible provided she completed her definitive anticancer treatment more than 3 years ago and she remains breast cancer disease free prior to start of study treatment.

E-5. Patient with myelodysplastic syndrome/acute myeloid leukemia history E-6. Patient having experienced for at least one cycle, a delay > 2 weeks due to prolonged hematological recovery during the first line chemotherapy E-7. Patient receiving radiotherapy within 6 weeks prior to study treatment E-8. Major surgery within 4 weeks of starting study treatment and patient must have recovered from any effects of any major surgery E-9. Previous allergenic bone marrow transplant. E-10. Any previous treatment with PARP inhibitor, including olaparib. E-11. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroidal antiemetics).

E-12. Current or recent (within 10 days prior to randomization) chronic use of aspirin > 325 mg/day.

E-13. Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.

E-14. Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.

E-15. Clinically significant (e.g. active) cardiovascular disease, including:

1. Myocardial infarction or unstable angina within ≤ 6 months of randomization,
2. New York Heart Association (NYHA) ≥ grade 2congestive heart failure (CHF).
3. Poorly controlled cardiac arrhythmia despite medication (patient with rate controlled atrial fibrillation are eligible), or any clinically significant abnormal finding on resting ECG,
4. Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision).

E-16. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub- Arachnoids Hemorrhage (SAH) within 6 months prior to randomization.

E-17. History or evidence of hemorrhagic disorders within 6 months prior to randomization.

E-18. Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation).

E-19. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of suspected spinal cord compression.

E-20. History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).

E-21. Significant traumatic injury during 4 weeks prior to randomization. E-22. Non-healing wound, active ulcer or bone fracture. Patient with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection is eligible but require 3 weekly wound examinations.

E-23. History of VEGF therapy related abdominal fistula or gastrointestinal perforation or active gastrointestinal bleeding within 6 months prior to the first study treatment.

E-24. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease.

E-25. Patient with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.

E-26. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.

E-27. Pregnant or lactating women. E-28. Participation in another clinical study with an investigational product during her chemotherapy course immediately prior to randomization.

E-29. Patient unable to swallow orally administered medication and patient with gastrointestinal disorders likely to interfere with absorption of the study medication.

E-30. Patient with a known hypersensitivity to olaparib or any of the recipients of the product.

E-31. Immunocompromised patient, e.g., with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids or patient who is known to be serologically positive for human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Efficacy by progression free survival (PFS1) | phase up to a total of 15 months

SECONDARY OUTCOMES:
Overall survival | Study end
  Overall survival is defined as the time from the date of randomization until death due to any cause.
Time to earliest progression by RECIST or CA-125 | Study end
  Time to earliest progression by RECIST v. 1.1 or CA-125 or death is defined as the time from randomization to the earliest date of RECIST or CA-125 progression or death by any cause.
Second Progression Free Survival (PFS2) | Study end
  Time from randomization to second progression is defined as the time from the date of randomization to the earliest of the progression event subsequent to that used for the primary variable PFS, or date of death.
Time to start of first subsequent therapy or death (TFST) | Study end
  Time to start of first subsequent therapy or death (TFST) will be assessed. TFST is defined as the time from the date of randomization to the earliest of the date of anti-cancer therapy start date following study treatment discontinuation, or death.
Time to start of second subsequent therapy or death (TSST) | Study end
  Time to start of second subsequent therapy or death (TSST) will be assessed. TSST is defined as the time from the date of randomization to the earliest of the date of second subsequent anti-cancer therapy start date following study treatment discontinuation, or death.
Safety and Tolerability | Study end
Patient reported outcome | 2 years after last patient included

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAY COQUARD, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (163):
- Austria (6):
  - KH der Barmherzigen Brüder Graz, Graz
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Landeskrankenhaus Salzburg, Salzburg
  - Medical University of Vienna, Vienna
  - Krankenhaus Hietzing, Vienna
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Gasthuisberg, Leuven
  - Hôpital de la Citadelle, Liège
  - Clinique et maternité Sainte Elisabeth, Namur
  - CHU Dinant Godinne, Yvoir
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
- Finland (4):
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (43):
  - Hôpital Européen Georges Pompidou, Paris, Ilhe de France
  - ICO Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Hôpital Michallon - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Huriez, Lille
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Catherine de Sienne - Group confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Institut Curie - Hopital Claudius Régaud, Paris
  - Hôpital des Diaconesses, Paris
  - Hôpital Cochin, Paris
  - Hopital Tenon, Paris
  - Groupe Hospitalier Saint-Joseph, Paris
  - Clinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - Hôpital de la Milétrie - CHU de Poitiers - Pôle Régional de Cancérologie, Poitiers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital René Huguenin, Institut Curie, Saint-Cloud
  - ICO Centre René Gauducheau, Saint-Herblain
  - Centre de Radiothérapie - Clinique Sainte-Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur - ONCOSUD, Toulouse
  - ICL Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (59):
  - Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Hochtaunus-Kliniken, Bad Homburg
  - Praxisklinik Krebsheilkunde für Frauen, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Charité - Universitätsmedizin Berlin (CVK), Berlin
  - Onkologie Bottrop, Bottrop
  - GYNAEKOLOGICUM Bremen, Bremen
  - Universitätsfrauenklinik Köln, Cologne
  - St. Elisabeth Krankenhaus, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsfrauenklinik Erlangen, Erlangen
  - Kliniken Essen Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt
  - Universitätsfrauenklinik Freiburg, Freiburg im Breisgau
  - Universitäts-Frauenklinik Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Klinkum Gütersloh, Gütersloh
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Albertinen Krankenhaus, Hamburg
  - Gynäkologisch-Onkologische Praxis Hannover, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - St. Vincentius Kliniken, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum Konstanz, Konstanz
  - HELIOS Klinikum Krefeld, Krefeld
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Johannes Wesling Klinikum, Minden
  - Klinikum der Universität München, München
  - Klinikum rechts der Isar, München
  - Universitätsklinikum Münster, Münster
  - Kliniken des Landkreises Neumarkt, Neumarkt
  - Sana Klinikum Offenbach, Offenbach
  - Ortenau Klinikum, Offenburg
  - Onkologie Ravensburg, Ravensburg
  - Universitätsfrauenklinik Regensburg, Regensburg
  - Klinikum am Steinenberg, Reutlingen
  - ROMed Klinikum Rosenheim, Rosenheim
  - Klinikum Südstadt, Rostock
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitäts-Frauenklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - HELIOS Dr. Horst Schmidt Kliniken, Wiesbaden
  - Marien Hospital Witten, Witten
  - amO Wolfsburg, Wolfsburg
  - Klinikum Worms, Worms
  - Universitätsklinikum Würzburg, Würzburg
- Italy (20):
  - Centro Riferimento Oncologico, Aviano
  - Policlinico S.Orsola-Malpighi, Bologna
  - Spedali Civili-Università di Brescia, Brescia
  - Ospedale Senatore Antonio Perrino, Brindisi
  - EO Ospedali Galliera, Genova
  - Ospedale San Luca, Lucca
  - Istituto Nazionale Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori - IRCCS Pascale, Napoli
  - Istituto Oncologico Veneto, Padua
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale Santa Chiara, Pisa
  - AO ASL 4 - Ospedale di Prato, Prato
  - Arcispedale S. M. Nuova, Reggio Emilia
  - Istituto Regina Elena, Roma
  - Policlinico Umberto I La Sapienza, Roma
  - Policlinico Universitario Gemelli Università Cattolica del Sacro Cuore, Roma
  - Ospedale S. Anna, Torino
  - Ospedale Mauriziano, Torino
  - Ospedale Santa Chiara, Trento
- Japan (7):
  - Ehime University Hospital, Ehime
  - Hyogo Cancer Center, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Kagoshima University Medical And Dental Hospital, Kagoshima
  - Saitama Medical University International Medical Center, Saitama
  - Jichi Medical University Hospital, Tochigi
  - National Cancer Center Hospital, Tokyo
- Centre Hospitalier Princesse Grace, Monaco, Monaco
- Spain (14):
  - H. U. Fundación Alcorcón, Alcorcón
  - H. de la Santa Creu i Sant Pau, Barcelona
  - C.S. Parc Taulí, Barcelona
  - H. U. Reina Sofía, Córdoba
  - H.U. Arnau de Vilanova, Lleida
  - MD Anderson Cancer Center Madrid, Madrid
  - H. U. Ramón y Cajal, Madrid
  - H. U. 12 de Octubre, Madrid
  - H.U. Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Instituto Valenciano de Oncología, Valencia
  - H. General Universitario de Valencia, Valencia
  - H. U. P. La Fe, Valencia
  - H. U. Miguel Servet, Zaragoza
- Linköping University Hospital, Linköping, Sweden

REFERENCES:
- [Result] Ray-Coquard I, Pautier P, Pignata S, Perol D, Gonzalez-Martin A, Berger R, Fujiwara K, Vergote I, Colombo N, Maenpaa J, Selle F, Sehouli J, Lorusso D, Guerra Alia EM, Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marme F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428. doi: 10.1056/NEJMoa1911361. PMID 31851799
- [Derived] Barnicle A, Ray-Coquard I, Rouleau E, Cadoo K, Simpkins F, Aghajanian C, Leary A, Poveda A, Lheureux S, Pujade-Lauraine E, You B, Ledermann J, Matulonis U, Gourley C, Timms KM, Lai Z, Hodgson DR, Elks CE, Dearden S, Egile C, Lao-Sirieix P, Harrington EA, Brown JS. Patterns of genomic instability in > 2000 patients with ovarian cancer across six clinical trials evaluating olaparib. Genome Med. 2024 Dec 18;16(1):145. doi: 10.1186/s13073-024-01413-5. PMID 39695768
- [Derived] Montegut C, Falandry C, Cinieri S, Cropet C, Montane L, Rousseau F, Joly F, Moubarak M, Mosconi AM, Guerra-Alia EM, Schauer C, Fujiwara H, Vergote I, Parma G, Lindahl G, Anota A, Canzler U, Marme F, Pujade-Lauraine E, Ray-Coquard I, Sabatier R. Safety and quality of life with maintenance olaparib plus bevacizumab in older patients with ovarian cancer: subgroup analysis of PAOLA-1/ENGOT-ov25. Oncologist. 2025 Jul 4;30(7):oyae322. doi: 10.1093/oncolo/oyae322. PMID 39673779
- [Derived] Harter P, Marth C, Mouret-Reynier MA, Cropet C, Lorusso D, Guerra-Alia EM, Matsumoto T, Vergote I, Colombo N, Maenpaa J, Lebreton C, de Gregorio N, Mosconi AM, Rubio-Perez MJ, Bourgeois H, Fasching PA, Cecere SC, Hardy-Bessard AC, Denschlag D, de Percin S, Hanker L, Favier L, Bauerschlag D, Desauw C, Hillemanns P, Largillier R, Sehouli J, Grenier J, Pujade-Lauraine E, Ray-Coquard I; PAOLA-1/ENGOT-ov25 investigators. Efficacy of subsequent therapies in patients with advanced ovarian cancer who relapse after first-line olaparib maintenance: results of the PAOLA-1/ENGOT-ov25 trial. Ann Oncol. 2025 Feb;36(2):185-196. doi: 10.1016/j.annonc.2024.10.828. Epub 2024 Nov 9. PMID 39528049
- [Derived] Lorusso D, Mouret-Reynier MA, Harter P, Cropet C, Caballero C, Wolfrum-Ristau P, Satoh T, Vergote I, Parma G, Nottrup TJ, Lebreton C, Fasching PA, Pisano C, Manso L, Bourgeois H, Runnebaum I, Zamagni C, Hardy-Bessard AC, Schnelzer A, Fabbro M, Schmalfeldt B, Berton D, Belau A, Lotz JP, Gropp-Meier M, Gladieff L, Luck HJ, Abadie-Lacourtoisie S, Pujade-Lauraine E, Ray-Coquard I. Updated progression-free survival and final overall survival with maintenance olaparib plus bevacizumab according to clinical risk in patients with newly diagnosed advanced ovarian cancer in the phase III PAOLA-1/ENGOT-ov25 trial. Int J Gynecol Cancer. 2024 Apr 1;34(4):550-558. doi: 10.1136/ijgc-2023-004995. PMID 38129136
- [Derived] Callens C, Rodrigues M, Briaux A, Frouin E, Eeckhoutte A, Pujade-Lauraine E, Renault V, Stoppa-Lyonnet D, Bieche I, Bataillon G, Karayan-Tapon L, Rochelle T, Heitz F, Cecere SC, Perez MJR, Grimm C, Nottrup TJ, Colombo N, Vergote I, Yonemori K, Ray-Coquard I, Stern MH, Popova T. Shallow whole genome sequencing approach to detect Homologous Recombination Deficiency in the PAOLA-1/ENGOT-OV25 phase-III trial. Oncogene. 2023 Nov;42(48):3556-3563. doi: 10.1038/s41388-023-02839-8. Epub 2023 Nov 9. PMID 37945748
- [Derived] Pujade-Lauraine E, Brown J, Barnicle A, Wessen J, Lao-Sirieix P, Criscione SW, du Bois A, Lorusso D, Romero I, Petru E, Yoshida H, Vergote I, Colombo N, Hietanen S, Provansal M, Schmalfeldt B, Pignata S, Martin Lorente C, Berton D, Runnebaum IB, Ray-Coquard I. Homologous Recombination Repair Gene Mutations to Predict Olaparib Plus Bevacizumab Efficacy in the First-Line Ovarian Cancer PAOLA-1/ENGOT-ov25 Trial. JCO Precis Oncol. 2023 Jan;7:e2200258. doi: 10.1200/PO.22.00258. PMID 36716415
- [Derived] Gonzalez-Martin A, Desauw C, Heitz F, Cropet C, Gargiulo P, Berger R, Ochi H, Vergote I, Colombo N, Mirza MR, Tazi Y, Canzler U, Zamagni C, Guerra-Alia EM, Levache CB, Marme F, Bazan F, de Gregorio N, Dohollou N, Fasching PA, Scambia G, Rubio-Perez MJ, Milenkova T, Costan C, Pautier P, Ray-Coquard I; PAOLA1/ENGOT-ov25 investigators. Maintenance olaparib plus bevacizumab in patients with newly diagnosed advanced high-grade ovarian cancer: Main analysis of second progression-free survival in the phase III PAOLA-1/ENGOT-ov25 trial. Eur J Cancer. 2022 Oct;174:221-231. doi: 10.1016/j.ejca.2022.07.022. Epub 2022 Sep 5. PMID 36067615
- [Derived] Fujiwara K, Fujiwara H, Yoshida H, Satoh T, Yonemori K, Nagao S, Matsumoto T, Kobayashi H, Bourgeois H, Harter P, Mosconi AM, Vazquez IP, Reinthaller A, Fujita T, Rowe P, Pujade-Lauraine E, Ray-Coquard I. Olaparib plus bevacizumab as maintenance therapy in patients with newly diagnosed, advanced ovarian cancer: Japan subset from the PAOLA-1/ENGOT-ov25 trial. J Gynecol Oncol. 2021 Sep;32(5):e82. doi: 10.3802/jgo.2021.32.e82. PMID 34378365
- See also: Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer — http://www.ncbi.nlm.nih.gov/pubmed/31851799